CLINICAL TRIAL: NCT06169995
Title: A Multi-center, Open-label，Single-arm Clinical Trial to Evaluate the Efficacy and Safety of Remimazolam Tosilate for Injection for Sedation in Upper Gastrointestinal Endoscopy
Brief Title: A Study of Remimazolam Tosilate for Sedation in the Upper Gastrointestinal Endoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR7056-402
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Sedation in the Upper Gastrointestinal Endoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remimazolam Tosilate for Injection (Experimental)
  Interventions: Drug: Remimazolam Tosilate

INTERVENTIONS:
Drug: Remimazolam Tosilate — bolus dose: 5mg，IV supplemental dose: 2.5mg，IV

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Remimazolam Tosilate for Injection for sedation in Upper Gastrointestinal Endoscopy

ELIGIBILITY:
Inclusion Criteria:

1. patients or their guardians are able to provide a written informed consent
2. participants undergo upper gastrointestinal endoscopy
3. ≥18 years old, male or female
4. 18 kg/m2≤bmi≤30kg/m2

Exclusion Criteria:

1. Subjects to be intubated (including laryngeal mask placement);
2. Complex endoscopic diagnosis and treatment operations are required;
3. Severe cardiovascular disease within 6 months prior to signing the ICF;
4. Heart rate < 50 beats/min during screening period;
5. Subjects with poor blood pressure control during screening;
6. Severe arrhythmias or heart disease; the circulatory system is unstable;
7. Subjects with a history of severe cardiovascular disease, or cerebrovascular disease, or neurological disease, or mental illness
8. Subjects with a history of drug abuse;
9. Abnormal values of the laboratory examination;
10. Allergic to relevant drugs ingredient or component;
11. Pregnant or nursing women;
12. Subjects who has participated in clinical trials of other interventions recently;
13. Other conditions deemed unsuitable to be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-12-11 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-16 (Actual)

PRIMARY OUTCOMES:
Percentage(%) of paticipants who experienced successful sedation in Upper Gastrointestinal Endoscopy | on Day1

SECONDARY OUTCOMES:
Percentage of subjects receiving supplemental dose for sedation | on Day1
The number of supplemental doses of the research drug | on Day1
Wake-up time. | on Day1
Incidence of sedation hypotension. | on Day1
Incidence of respiratory depression | on Day1

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Affiliated Hospital Of Guizhou Medical University, Guiyang, Guizhou
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided